CLINICAL TRIAL: NCT07163676
Title: Is There a Response of Glaucoma to Baduanjin Exercise in Elders?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of physical therapy for Cardiovascular, Respiratory disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00014233-35
Record Dates: First submitted 2025-09-02; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group number 1 (Experimental): group I will receive baduanjin exercise for 60 minutes every day ((except fridays) for eight weeks.
  Interventions: Behavioral: Baduanjin exercise
- group number 2 (No Intervention): group II will act as waistlist.

INTERVENTIONS:
Behavioral: Baduanjin exercise — group I will receive baduanjin exercise for 60 minutes every day ((except fridays) for eight weeks.
  Arms: group number 1

SUMMARY:
glaucoma is prevalent between elders. Baduanjin exercise is a suitable exercise for elders. elders with glaucoma will divided to group I or group II. each/every group will contain 30 elders. group I will receive baduanjin exercise for 60 minutes every day ((except fridays) for eight weeks. group II will act as waistlist.

DETAILED DESCRIPTION:
Baduanjin exercise is a suitable exercise for elders. elders with glaucoma will divided to group I or group II. each/every group will contain 30 elders. group I will receive baduanjin exercise for 60 minutes every day ((except fridays) for eight weeks. group II will act as waistlist.

ELIGIBILITY:
Inclusion Criteria:

* high-tension primary open angle glaucoma (bilateral)
* ocular hypertension in both eyes

Exclusion Criteria:

* cataract
* diabetes
* cardiac disorders
* obesity

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — based on self-representation of gender identity.
Enrollment: 60 (Estimated)
Dates: Start 2025-05-11 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
intraocular pressure | it will be measured after 8 weeks
  it will be assessed in both eyes

SECONDARY OUTCOMES:
patient health questionnaire | it will be measured after 8 weeks
  it is nine-item questionnaire assessing depression
National Eye Institute Visual Function Questionnaire | it will be measured after 8 weeks
  it is 25-item questionnaire
Glaucoma-related quality of life questionnaire | it will be measured after 8 weeks
  it is a quality of life questionnaire
State trait anxiety inventory | it will be measured after 8 weeks
  it is a questionnaire about anxiety
Stress vulnerability scale | it will be measured after 8 weeks
  it is a questionnaire about Stress vulnerability

CONTACTS AND LOCATIONS:
Overall Officials: Ali MA Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Giza, Dokki, Egypt